CLINICAL TRIAL: NCT03026036
Title: Neuroimaging Studies of Reward Processing in Depression
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2015P002520
Record Dates: First submitted 2016-12-27; First posted 2017-01-20 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression; MRI; PET; Reward
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Magnetic Resonance Spectroscopy; Raclopride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples, saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MDD: Patients with current Major Depressive Disorder
  Interventions: Radiation: PET Scan with Raclopride
- rMDD: Patients with a history of Major Depressive Disorder
  Interventions: Radiation: PET Scan with Raclopride
- HC: Healthy control participants
  Interventions: Radiation: PET Scan with Raclopride

INTERVENTIONS:
Radiation: PET Scan with Raclopride — A subsample (21 per group) will complete the PET imaging.

SUMMARY:
This study investigates stress-related signaling of glutamate and dopamine within the reward-processing circuit in Major Depressive Disorder (MDD), and whether they can be used to predict depressive symptoms in the future. This will be achieved through various neuroimaging tools (MRS, fMRI, PET), behavioral tasks, and a naturalistic follow-up design.

DETAILED DESCRIPTION:
The overarching goals of this research are to investigate: (1) stress-induced glutamatergic abnormalities and their relation to disruption within the corticostriatal valuation circuit in MDD; (2) stress-induced DA signaling disruptions in MDD; and (3) the predictive validity of these two pathophysiological mechanisms. This will be achieved through an innovative integration of (1) proton magnetic resonance spectroscopy (MRS)-based assessments of glutamatergic metabolites in the mPFC; (2) functional magnetic resonance imaging (fMRI) probes of the corticostriatal valuation circuit with well-established stress manipulations (MAST) and assessments (cortisol and inflammatory markers); (3) positron emission tomography (PET)-based measurement of striatal DA release with well-established stress manipulations and assessments (cortisol and inflammatory markers); and (4) a naturalistic follow-up design.

ELIGIBILITY:
General Inclusion Criteria:

* All genders, races, and ethnic origins, aged between 18 and 45
* Capable of providing written informed consent, and fluent in English
* Right-handed
* Absence of any psychotropic medications for at least 2 weeks

Inclusion Criteria for Current Depression Group (MDD):

* Current DSM-5 diagnostic criteria for MDD (as diagnosed with the use of the SCID)

Inclusion Criteria for Remitted Depression Group (rMDD):

* History of at least one major depressive episode within the past five years
* Not currently depressed

Inclusion Criteria for Healthy Control Group (HC):

* Absence of any medical, neurological, and psychiatric illness (including alcohol/substance abuse)

Exclusion Criteria:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician
* Pregnant women
* Failure to meet standard MRI or PET safety requirements
* Serious or unstable medical illness
* History of seizure disorder
* History or current diagnosis of organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, OCD, PTSD, mood congruent or mood incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of cocaine or stimulant abuse, which will lead to automatic exclusion)
* Simple phobia, social anxiety disorder, and generalized anxiety disorder will be allowed only if secondary to MDD and only in the MDD group
* History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine)
* History of use of dopaminergic drugs (including methylphenidate)
* Patients with a lifetime history of electroconvulsive therapy (ECT)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current Major Depressive Disorder (MDD), or Remitted Major Depressive Disorder (rMDD)
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Behavioral Performance on the Probabilistic Stimulus Selection Task | Screening visit (Day 0)
  The Probablilistic Reward Task operationalizes positive reinforcement learning
MRI Data | MRI scans for a total of 90 minutes take place within 30 days of Screening Visit
PET scan with raclopride | a total of 90 minutes take place after the MRI data collection
Salivary Cortisol | 6 times during MRI visit (on or before Day 30), and 4 times during PET visit (on or before Day 30)
Four Blood Samples (6ml) | During the MRI visit (on or before Day 30)
Follow-up Clinical Interviews | 6 months and 12 months after the MRI scanning visit
Behavioral Performance on the Instrumental Learning Task | Administered during MRI scan (on or before Day 30)
  The instrumental learning task is designed to measure participant learning from reward and punishment.

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- David Crowley, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared via NIMH Data Archive (as part of data submission agreement)
Time Frame: All collected IPD are shared every 6 months (1/15 and 7/15 of each year)
Access Criteria: Investigators may request for access for approval by the NIMH.